CLINICAL TRIAL: NCT00957450
Title: Validation Study of Modeled Intra-pelvic Organ Motion During External Beam Radiotherapy for Cervix Cancer Using Frequent Magnetic Resonance Imaging
Brief Title: Intra-Pelvic Organ Motion for Cervix Cancer Patient Using Imaging
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: UHN REB 08-0043-CE
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Cervix Cancer
Keywords: cervix cancer; intra-pelvic organ motion; cervical cancer and CBCT
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Impact of organ motion
  Characterize the impact of normal organ motion in the pelvic on tumour movement, during treatment. This will be assessed in patients with pelvic cancer.

SUMMARY:
Patients with cervix cancer having radiotherapy experience side-effects because the radiotherapy fields have to be quite large to account for tumour movement in the pelvis during treatment, this irradiates a lot of normal tissues. This study aims to characterize and model the tumour motion, as well as the motion of surrounding normal tissues, during treatment. By doing this, the investigators can look at ways to minimise tumour motion and spare more normal tissues. By tailoring the radiotherapy dose more accurately, the investigators will reduce the side-effects of treatment and improve local control of the tumour. By doing multiple magnetic resonance imaging (MRI) scans of the patients during treatment, the investigators can identify where the tumour and surrounding normal tissues are at that point in time. Collecting all the information from these scans, will allow the investigators to model the motion of the tumour and these pelvic organs, and investigate the best way to target the tumour while still sparing normal tissues.

DETAILED DESCRIPTION:
At simulation: patients will have two MRI scans in addition to the standard planning CT scan. One MRI scan will be with bladder full, the other will be with bladder empty. During treatment: patients will have two or three MRI scans per week at their convenience. MRI scans will be scheduled close to radiotherapy treatment times to minimise inconvenience for the patient. On the same day they have an MRI scan, they will also have a CBCT at the time of treatment. None of the images will be used to alter or influence the treatment the patient is receiving. If the patient feels that the imaging schedule is too inconvenient, they will be given the option to reduce the frequency of the scanning or to withdraw from the study.All the images will be loaded onto a password secure server. The MRI scans will be fused to the planning CT scan using bone-to-bone matching. Tumour and intra-pelvic organs will be contoured on the MRI scans. The contours will be used to create surface meshes of each organ and with research software, we will be able to model the motion and deformation of these organs over the course of radiotherapy. Using this data, we will be able to simulate the dose impact of the organ motion on different intensity-modulated radiotherapy plans. We will also explore the impact of bladder & rectal filling on tumour motion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18years
* Biopsy confirmed cervix cancer
* Not suitable for surgery
* Suitable for radical radiotherapy
* ECOG 0-2
* Informed consent

Exclusion Criteria:

* Patients unwilling or unable to give informed consent
* Prior pelvic radiotherapy
* Contraindications to MRI scan

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, the organ motion of Patients with cervical cancer will be assessed. The study population will be selected from clinic.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-02; Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Measure inter-fraction organ movements associated with cervix cancer during the course of definitive radiotherapy. Characterise the impact of bladder and rectal filling on target motion during a course of definitive radiotherapy | 24 months

SECONDARY OUTCOMES:
Model intra-pelvic organ motion during RT. Model tumour & normal tissue dose accumulation. Perform planning studies on the image data sets. Investigate the utility of tumour localisation surrogates using CBCT & MR imaging. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Milosevic, MD, Principal Investigator — Univesity Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Toronto, Ontario, Canada